CLINICAL TRIAL: NCT02482870
Title: Comparison of King Vision Video Laryngoscope and Macintosh Laryngoscope in Terms of First Pass Intubation Success Rate, Intubation Time, Glottic View Time, and Complications Related to Laryngoscopy
Brief Title: Efficiency of the King Vision Video Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Başar Erdivanlı, Asst Prof, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 2014/109
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Respiratory Failure; Intubation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Patients scheduled for general anesthesia with endotracheal intubation will be randomized to either intubation with Macintosh laryngoscope first or King Vision videolaryngoscope first. All patients will be intubated with both laryngoscopes.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Macintosh (Active Comparator): Patients scheduled for general anesthesia during the study period, who had been intubated with Macintosh laryngoscope first and then with KingVision videolaryngoscope.
  Interventions: Device: Macintosh laryngoscope; Device: King Vision video laryngoscope
- KingVision (Active Comparator): Patients scheduled for general anesthesia during the study period, who had been intubated with King Vision videolaryngoscope first and then with Macintosh laryngoscope.
  Interventions: Device: Macintosh laryngoscope; Device: King Vision video laryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope — Using a Macintosh laryngoscope, time to glottic view, best Cormack-Lehane grade, time to intubation, time to first ventilation has been recorded.
Device: King Vision video laryngoscope — Using a King Vision video laryngoscope, time to glottic view, best Cormack-Lehane grade, time to intubation, time to first ventilation has been recorded.

SUMMARY:
The investigators studied the efficiency of Macintosh laryngoscope and the King Vision video laryngoscope in adult patients scheduled for general anesthesia. Best Cormack-Lehane score obtained, glottic view time, intubation time, time to ventilation, correlation between the Mallampati classification and the Cormack-Lehane grades, and complications related to laryngoscopy and intubation has been investigated.

DETAILED DESCRIPTION:
Securing the airway is essential in general anesthesia. Anesthetic problems related to airway management constitute 17% of closed claims, difficult intubation being the most common one with an occurrence rate of 5%. Problems like delayed intubation, misplaced tracheal tube, or airway trauma are frequently seen in outpatient settings and end up with either death or hypoxic brain damage. Therefore, preoperative visit should include detailed assessment of the airways according to clues of difficult intubation.Several studies compared the King Vision video laryngoscope with other laryngoscopes in manikins simulating difficult airway scenarios, and reported better glottic views. The investigators aimed to study the correlation between the Mallampati classification and the glottic views (Cormack-Lehane grade) obtained with Macintosh laryngoscopy, and the King Vision video laryngoscopy in adult patients scheduled for general anesthesia. Secondary outcomes will be successful intubation rate, time to obtain the best view, time to successful intubation, and complications related to laryngoscopy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for general anesthesia
* age higher than 18 years
* age lower than 60 years

Exclusion Criteria:

* emergency surgery
* mouth opening less than 2 cm
* American Society of Anesthesiologists (ASA) score higher than 2
* oropharyngeal anomaly
* glottic or supraglottic mass
* history of surgery due to oropharyngeal anomaly, glottic or supraglottic mass

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 388 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Başar Erdivanli, Asst. Prof., Principal Investigator — Recep Tayyip Erdogan Univeristy, Medical Faculty, Department of Anesthesiology and Reanimation
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Metzner J, Posner KL, Lam MS, Domino KB. Closed claims' analysis. Best Pract Res Clin Anaesthesiol. 2011 Jun;25(2):263-76. doi: 10.1016/j.bpa.2011.02.007. PMID 21550550
- [Background] Woodall NM, Benger JR, Harper JS, Cook TM. Airway management complications during anaesthesia, in intensive care units and in emergency departments in the UK". Trends in Anaesthesia and Critical Care 2(2): 58-64, 2012.
- [Background] Yentis SM. Predicting difficult intubation--worthwhile exercise or pointless ritual? Anaesthesia. 2002 Feb;57(2):105-9. doi: 10.1046/j.0003-2409.2001.02515.x. No abstract available. PMID 11871945
- [Background] Akihisa Y, Maruyama K, Koyama Y, Yamada R, Ogura A, Andoh T. Comparison of intubation performance between the King Vision and Macintosh laryngoscopes in novice personnel: a randomized, crossover manikin study. J Anesth. 2014 Feb;28(1):51-7. doi: 10.1007/s00540-013-1666-9. Epub 2013 Jun 30. PMID 23812581
- [Background] Murphy LD, Kovacs GJ, Reardon PM, Law JA. Comparison of the king vision video laryngoscope with the macintosh laryngoscope. J Emerg Med. 2014 Aug;47(2):239-46. doi: 10.1016/j.jemermed.2014.02.008. Epub 2014 Apr 16. PMID 24742495
- [Background] Yun BJ, Brown CA 3rd, Grazioso CJ, Pozner CN, Raja AS. Comparison of video, optical, and direct laryngoscopy by experienced tactical paramedics. Prehosp Emerg Care. 2014 Jul-Sep;18(3):442-5. doi: 10.3109/10903127.2013.864356. Epub 2014 Jan 24. PMID 24460509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adult patients scheduled for general anesthesia with intubation in Recep Tayyip Erdogan University Education and Research Hospital. The last patient completed in July 2014.
Pre-assignment Details: None of the 388 patients enrolled between January 2014 and July 2014 were excluded from the trial.
Groups:
- Macintosh First, Then King Vision: The patients has been intubated first with a Macintosh, then with a King Vision video laryngoscope.
- King Vision First, Then Macintosh: The patients has been intubated first with a King Vision video laryngoscope, then with a Macintosh laryngoscope.
Period: Overall Study
Arm/Group | Macintosh First, Then King Vision | King Vision First, Then Macintosh
Started (Period 1 started with the patient enrollment on 01.01.2014.) | 186 | 202
Completed (Period 1 ended on 21.01.2014.) | 186 | 202
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult patients scheduled for general anesthesia with endotracheal intubation.
Groups:
- All Study Participants: Each patient were intubated with both Macintosh and King Vision video laryngoscope sequentially. The order of the laryngoscopes was randomized by flipping a coin.
Arm/Group | All Study Participants
Number analyzed (Participants) | 388
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48.5 [37 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 230
Height, Continuous [Median (Inter-Quartile Range); unit: cm] | 171 [165 to 175]
Weight, Continuous [Median (Inter-Quartile Range); unit: kg] | 80 [70 to 88]
Body mass index, Continuous [Median (Inter-Quartile Range); unit: kg/m^2] | 26.9 [24.3 to 30.9]
History of obstructive sleep apnea, Categorical [Count of Participants; unit: Participants]
  0 - No history of obstructive sleep apnea | 292
  1 - History of obstructive sleep apnea | 96
History of snoring, Categorical [Count of Participants; unit: Participants]
  0 - No history of snoring | 246
  1 - History of snoring | 142
Mallampati class, Categorical [Count of Participants; unit: Participants] — Mallampati class is used to indirectly assess the distance between the base of the tongue and the roof of the mouth, to predict how difficult an intubation will be.
  Participants
    0 - Ability to see any part of the epiglottis | 0
    1 - Soft palate, fauces, uvula, pillars visible | 79
    2 - Soft palate, fauces, uvula visible | 113
    3 - Soft palate, base of uvula visible | 107
    4 - Soft palate not visible at all | 89
American Society of Anesthesiologists score, Categorical [Count of Participants; unit: Participants] — "American Society of Anesthesiologists score" is a widely used grading system for preoperative health of the surgical patients.
  It is based on five classes (I to V):
  I-a completely healthy fit patient.
  II-patient has mild systemic disease.
  III-patient has severe systemic disease that is not incapacitating.
  IV-patient has incapacitating disease that is a constant threat to life.
  V-a moribund patient, not expected to live 24 hour w/out surgery. E-designates emergency surgery (added after roman literal like "IIE").
  Participants
    1 - A normal healthy patient | 192
    2 - A patient with mild systemic disease | 196
Thyromental distance, Continuous [Median (Inter-Quartile Range); unit: cm] | 6.2 [5.3 to 7.3]
Sternomental distance, Continuous [Median (Inter-Quartile Range); unit: cm] | 10.9 [9.6 to 12.3]
Interincisor distance, Continuous [Median (Inter-Quartile Range); unit: cm] | 3.3 [2.7 to 4.1]

OUTCOME MEASURES:

1. Primary Outcome: Intubation Success Rate
Description: Endotracheal intubation attempt is defined as entrance of the endotracheal tube into the patient's mouth. Any major change in the alignment of the laryngoscope is defined as another intubation attempt. Successful endotracheal intubation is defined as the endotracheal cuff passing through the patient's vocal cords. Intubation success rate is defined as: 1 / [the number of attempts].
Time Frame: less than 24 hours
Measure: Number; unit: participants
Groups:
- Macintosh: Using a Macintosh laryngoscope, first pass intubation success rate has been recorded.
- King Vision Video Laryngoscope: Using a King Vision video laryngoscope, first pass intubation success rate has been recorded.
Arm/Group | Macintosh | King Vision Video Laryngoscope
Number analyzed (Participants) | 388 | 388
participants
  0 - Could not be intubated | 22 | 13
  1 - Successfully intubated | 366 | 375
Statistical Analysis 1: Comparison: Macintosh vs King Vision Video Laryngoscope; Sample size was calculated according to the first 60 patients. To obtain 90% power with an alpha error of 0.05, a total of 378 patients were required. Considering a possible drop-out rate of 2.5% due to unexpected complications, we aimed for 388 patients; Test type: Superiority or Other; p = 0.119, Chi-squared — A priori threshold for statistical significance was 0.05; Chi-square value = 2.424; degrees of freedom = 1

2. Secondary Outcome: Intubation Time
Description: Successful endotracheal intubation is defined as the endotracheal cuff passing the patient's vocal cords. Time to intubation with each laryngoscope is recorded.
Time Frame: less than 24 hours
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Macintosh: Using a Macintosh laryngoscope, intubation time has been recorded.
- King Vision Video Laryngoscope: Using a King Vision video laryngoscope, intubation time has been recorded.
Arm/Group | Macintosh | King Vision Video Laryngoscope
Number analyzed (Participants) | 388 | 388
seconds | 6.6 [5 to 8.9] | 10.8 [6.7 to 17.4]
Statistical Analysis 1: Comparison: Macintosh vs King Vision Video Laryngoscope; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [3 to 4.6]

3. Secondary Outcome: Glottic View Time
Description: Glottic view time (as defined when the laryngoscopist declared the best Cormack-Lehane score) with each laryngoscope is recorded.
  Cormack-Lehane score is obtained by directly assessing the distance between the base of the tongue and the roof of the mouth to predict how difficult an intubation will be.
  It consists of 4 grades:
  1. full view of glottis (difficult intubation unlikely)
  2. partial view of glottis (~5% risk of difficult intubation)
  3. partial view of epiglottis, none of glottis seen (~90% risk of difficult intubation)
  4. neither glottis nor epiglottis seen (difficult intubation very likely)
Time Frame: less than 24 hours
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Macintosh: Using a Macintosh laryngoscope, glottic view time has been recorded.
- King Vision Video Laryngoscope: Using a King Vision video laryngoscope, glottic view time has been recorded.
Arm/Group | Macintosh | King Vision Video Laryngoscope
Number analyzed (Participants) | 388 | 388
seconds | 7.3 [5.8 to 8.8] | 7.9 [6 to 11.8]
Statistical Analysis 1: Comparison: Macintosh vs King Vision Video Laryngoscope; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance was 0.05; Mean Difference (Net) = 0.9, 95% CI 2-sided [0.5 to 1.4]

4. Secondary Outcome: Cormack-Lehane Score
Description: Best Cormack-Lehane score (as declared by the laryngoscopist) obtained with both laryngoscopes is recorded.
  Cormack-Lehane score is graded according to the following criteria (1 is best, and 4 is worst):
  1. full view of glottis (difficult intubation unlikely)
  2. partial view of glottis (~5% risk of difficult intubation)
  3. partial view of epiglottis, none of glottis seen (~90% risk of difficult intubation)
  4. neither glottis nor epiglottis seen (difficult intubation very likely)
Time Frame: less than 24 hours
Measure: Number; unit: participants
Groups:
- Macintosh: Using a Macintosh laryngoscope, best Cormack-Lehane score obtained has been recorded.
- King Vision Video Laryngoscope: Using a King Vision video laryngoscope, best Cormack-Lehane score obtained has been recorded.
Arm/Group | Macintosh | King Vision Video Laryngoscope
Number analyzed (Participants) | 388 | 388
participants
  1 - Most of the glottis is visible | 149 | 357
  2 - At most half of the glottis is seen | 139 | 31
  3 - Only the epiglottis is visible | 93 | 0
  4 - No laryngeal structures are visible | 7 | 0
Statistical Analysis 1: Comparison: Macintosh vs King Vision Video Laryngoscope; For each patient, the difference between Cormack-Lehane score and Mallampati class was calculated for each laryngoscope. As an example, the first patient had a Mallampati score 3. Macintosh laryngoscope provided a Cormack-Lehane score of 2, therefore the difference is - 1, calculated as "2 - 3". In the same patient, King Vision video laryngoscope provided a Cormack-Lehane score of 1, therefore the difference is - 2, calculated as "1 - 3". T-test was used to compare the differences; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — A priori threshold for statistical significance was 0.05; t value = -11.224, degrees of freedom = 773.99; Mean Difference (Net) = -0.81, 95% CI 2-sided [-0.95 to -0.67]

5. Secondary Outcome: Airway Complications
Description: Any complication related to the laryngoscopy and intubation, such as cut, bleeding, damage to the teeth, laryngospasm, bronchospasm, desaturation below 90%, is recorded.
Time Frame: The participants' will be followed for the duration of hospital stay, an expected average of 2 days
Measure: Number; unit: participants
Groups:
- Macintosh: Airway complications related to the use of Macintosh laryngoscope has been recorded.
- King Vision Video Laryngoscope: Airway complications related to the use of King Vision video laryngoscope has been recorded.
Arm/Group | Macintosh | King Vision Video Laryngoscope
Number analyzed (Participants) | 388 | 388
participants
  0 - No complication | 384 | 382
  1 - Minor cuts on the lips | 4 | 6
Statistical Analysis 1: Comparison: Macintosh vs King Vision Video Laryngoscope; Test type: Superiority or Other; p = 0.75, Chi-squared, Corrected — A priori threshold for statistical significance was 0.05; Chi-square test with Yates' continuity correction: chi-square = 0.101; degrees of freedom = 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Patients were supervised and observed for adverse events during the period they spent in the operating room, and post anesthetic care unit, by the attending anesthesiologist and anesthesia technician.
Groups:
- King Vision First, Then Macintosh: These patients had been intubated with a King Vision video laryngoscope first, and then with a Macintosh laryngoscope. Airway complications related to the laryngoscopy and intubation (cuts, bleeding, damage to the teeth, laryngospasm, bronchospasm, desaturation below 90%) had been recorded.
- Macintosh First, Then King Vision: These patients had been intubated with a Macintosh laryngoscope first, and then with a King Vision video laryngoscope. Airway complications related to the laryngoscopy and intubation (cuts, bleeding, damage to the teeth, laryngospasm, bronchospasm, desaturation below 90%) had been recorded.
Arm/Group | King Vision First, Then Macintosh | Macintosh First, Then King Vision
All-Cause Mortality (participants affected / at risk) | 6/202 | 4/186
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/186
Other Adverse Events (participants affected / at risk) | 3/202 | 3/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | King Vision First, Then Macintosh (N=202) | Macintosh First, Then King Vision (N=186)
Situation of "can't intubate, can't ventilate" (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Laryngospasm/Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Desaturation below 90% (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) — Fall of saturation of peripheral oxygen below 90%
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | King Vision First, Then Macintosh (N=202) | Macintosh First, Then King Vision (N=186)
Cuts on lips (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) — Minor cuts on lips occurring due to manipulations and pressure of the laryngoscope, mostly the blade.
Dental damage (Surgical and medical procedures) | 0 (0) | 0 (0) — Any kind of dental damage, such as enamel fracture or avulsion during laryngoscopy, were recorded.
Sore throat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) — Any case of painful or swollen throat were questioned at the entrance to and exit from the postanesthetic care unit by the anesthesia technician, and in the surgical ward by the nurse.

LIMITATIONS AND CAVEATS:
Sample size estimation according to small number of participants; sequential intubation with both laryngoscopes providing an advantage to the second laryngoscope.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes